CLINICAL TRIAL: NCT05099367
Title: Prostacyclin (PGI2) Pathway to Enhance Wound Healing in Diabetic Foot Ulcers
Acronym: PGI2HEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC18.314
Record Dates: First submitted 2021-10-04; First posted 2021-10-29 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Foot
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, pathophysiological study, comparing 3 parallel groups: healthy controls; patients with diabetes and without DFU; patients with diabetes and with DFU. To address secondary objectives , samples from a fourth group (patients with diabetes, neuropathy and DFU undergoing lower-limb amputation) will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 : healthy subject (Other): 15 healthy subject without diabetes
  Interventions: Diagnostic Test: Microdialysis, current induced vasodilation; Diagnostic Test: Skin biopsy
- Group 2 : diabetes without ulcer (Other): 15 patients with diabetes type II and without foot ulcer
  Interventions: Diagnostic Test: Microdialysis, current induced vasodilation; Diagnostic Test: Skin biopsy
- Group 3 : diabetes with ulcer active or <2 years (Other): 15 patients with diabetes type II and with foot ulcer (active or <2years)
  Interventions: Diagnostic Test: Microdialysis, current induced vasodilation; Diagnostic Test: Skin biopsy
- Group 4 : Patients with type 2 diabetes, neuropathy and DFU undergoing lower limb (Other): Patients with type 2 diabetes and neuropathy and DFU undergoing lower lunb surgery for skin ulcer
  Interventions: Diagnostic Test: peri-ulcerated skin biopsy

INTERVENTIONS:
Diagnostic Test: Microdialysis, current induced vasodilation — CIV will be applied over all microdialysis fibers: one perfused with saline, one perfused with a preferential COX-1 blocker; and one perfused with a preferential COX-2 blocker.
  CIV will be applied over all fibers in the following conditions: one perfused with saline, one perfused with fluconazole and L-NMMA, and the last one perfused with lidocaine.Dialysate collection will be performed after each CIV: dermal PGI2 metabolite (6-ketoPGF1α) and other COX-dependent prostanoids or metabolite (e.g. 11-dehydroTXB2) will be collected in the dialysate fluid and quantified. One hour after the last condition, treprostinil will be perfused over all fibers.
  Arms: Group 1 : healthy subject; Group 2 : diabetes without ulcer; Group 3 : diabetes with ulcer active or <2 years
Diagnostic Test: Skin biopsy — Skin biopsy will be proposed. It will be performed on the internal superior calf (medial gastrocnemius), at a reasonable distance from the foot
  Arms: Group 1 : healthy subject; Group 2 : diabetes without ulcer; Group 3 : diabetes with ulcer active or <2 years
Diagnostic Test: peri-ulcerated skin biopsy — Non-ulcerated skin from the peri-wound area will be collected. These patient will not undergo all the procedures included in this protocol.
  Arms: Group 4 : Patients with type 2 diabetes, neuropathy and DFU undergoing lower limb

SUMMARY:
Prospective, monocentric, pathophysiological study, comparing 3 parallel groups: healthy controls; patients with diabetes and without DFU; patients with diabetes and with DFU. To address secondary objectives, samples from a fourth group will be collected.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFUs) are a common and serious complication of diabetes mellitus, and associated with major morbidity. Indeed, diabetes is the primary cause of non-traumatic lower-limb amputation, and the rise in the prevalence of type 2 diabetes worldwide increases the global burden of DFUs. The treatment of DFUs is particularly challenging. Besides etiologic measures, local therapy of foot ulcers mainly relies on debridement of the wound and dressings. Essential complementary measures include pressure off-loading and infection control. However, despite these treatments, complications are frequent, stressing the need for new treatments.

The microcirculation has a key role in tissue survival, and several classical pathways explain how hyperglycemia damages the microvessels. There is growing evidence that the PGI2 pathway is dysregulated in diabetes, which contributes to microvascular dysfunction. Besides its vasodilator effect, recent data has revealed the major role of PGI2 in angiogenesis. In the skin, such effect on healing might be enhanced by the role of PGI2 in the regulation of fibroblast and keratinocytes migration and proliferation.

In the past few decades, studies in diabetic patients with ulcers have shown numerous structural and functional abnormalities of the cutaneous microcirculation, supporting its critical role in the pathophysiology of DFUs. However, the detailed mechanisms underlying endothelial dysfunction in the skin of diabetic patients remain largely unexplored in vivo. A better understanding of the specificities of microvascular changes in the diabetic foot is essential to developing new treatments for this pressing clinical need.

Objectives are

* to explore the role of the PGI2 pathway in skin microvascular reactivity, in healthy subjects and in diabetic patients with and without DFU
* To determine the involvement of COX-1 and COX-2 in cutaneous current-induced vasodilation (CIV), in healthy subjects and in diabetic patients with and without DFU.
* To determine the involvement of sensory nerves in cutaneous CIV, in healthy subjects and in diabetic patients with and without DFU.
* To compare the function of the IP receptor between healthy subjects and diabetic patients with and without DFU.
* To determine the involvement of the nitric oxide (NO) and epoxyeicosatrienoic acids (EETs) pathway in cutaneous CIV, in healthy subjects and in diabetic patients with and without DFU.
* To assess cutaneous expression of the different components of the PGI2 pathway in the skin of healthy subjects and of diabetic patients with and without DFU.
* To assess the role of the PGI2 pathway on cell migration in vitro

ELIGIBILITY:
Inclusion criteria:

Groups 1,2,3,4:

* Informed consent signed
* Affiliated to social security insurance or beneficiary of social security insurance
* Aged of 18 or older

Group 1: healthy volunteers:

-Free from all acute and chronic pathology

Group 2: diabetic patients without DFU:

-Patients with type 2 diabetes according to the criteria of the American Diabetes Association (ADA), without DFU or history of DFU

Group 3: diabetic patients with DFU or recent history of DFU (occurred within the last two years):

-Patients with type 2 diabetes according to the criteria of the American Diabetes Association (ADA) with: One or more active grade 1A, 1C, 2A or 2C (University of Texas Classification of Diabetic Foot) foot ulcer of microvascular or mixed etiology; Or a recent history (<2 years) of foot ulcer of microvascular or mixed etiology.

Group 4 (to collect samples of foot skin biopsies to address secondary objectives ):

-Patients with type 2 diabetes according to the criteria of the American Diabetes Association (ADA),with neuropathy and DFU undergoing lower-limb surgery for skin ulcer (e.g. toe amputation).

Exclusion criteria

Groups 1, 2 and 3:

* Unstable diabetes that has resulted in hyperosmolar coma or ketoacidosis, and/or documented increase or decrease in HbA1c of more than 2.0% within the previous 3 months.
* Presence of diabetic peripheral neuropathy above the ankle, defined as a scoring >3 of at least two of the four stimuli of the Neuropathy Disability Score (i.e. pinprick sensation, light touch, vibration, and temperature perception) (37).
* Infected wound, treated with antibiotics in the past 15 days.
* Critical ischemia of the lower limb, defined as leg pain at rest associated with ankle pressure <70 mmHg.
* History of hypersensitivity reaction to treprostinil, fluconazole, other azole compounds, L-NMMA, ketorolac, meloxicam, or any NSAIDs or acetylsalicylic acid, lidocaine (or any local anesthetic with an amide bond), or their excipients
* History of asthma, rhinitis, nasal polyps, angioedema, hives rash, or any other allergic reaction due to acetylsalicylic acid or any NSAID taking
* Pulmonary veno-occlusive disease (PVOD)
* Porphyria
* Hyperkalemia
* Active or uncontrolled cardiovascular disease as follows: Myocardial infarction, or angina within the previous 6 months; Severe ischemic heart disease; Arrhythmia (uncontrolled, symptomatic, requiring treatment or life-threatening); Congestive heart failure, or decompensated heart failure not medically controlled; Stroke or transient ischemic attack within the previous 3 months; Uncontrolled hypertension: systolic blood pressure (SBP)> 180 mmHg or diastolic blood pressure (DBP)> 105 mmHg (2 abnormal readings during visit) Valvular heart disease
* Severe liver disease (Child-Pugh C) at the time of enrollment
* Renal disease (creatinine >2 mg/dL and/or estimated glomerular filtration rate (GFR) <30 mL/min, history of dialysis)
* Active peptic ulcer disease, recent gastrointestinal bleeding or perforation, or history of peptic ulcer disease or gastrointestinal bleeding or perforation with NSAIDs
* Intracerebral or gastrointestinal hemorrhage, hemostasis disorder or every clinical status that may lead to bleeding
* Chronic venous disease defined as stage 4a and 4b of the Clinical-Etiological-Anatomical-Pathophysiological (CEAP) classification
* Cutaneous condition deemed incompatible with skin biopsy and dermal microdialysis by the investigator
* History of necrotic angiodermatitis
* Trauma or any clinical event susceptible to be responsible for hemorrhage within the previous 6 months
* Concomitant treatment with pentoxifylline, anticoagulants, probenecid, medicinal products known to prolong the QT interval or anti-inflammatory or analgesic dose of acetylsalicylic acid
* If concomitant treatment with NSAIDs, participants have to be stopped 1 week before the inclusion
* Pregnancy or Lactation
* Females with childbearing potential, defined as a premenopausal female capable of becoming pregnant, and not using an highly effective form of birth control. Effective birth control methods include: oral, implant or patch hormone contraception; intrauterine device; abstinence and outercourse; tubal ligation; vasectomy.

Groups 1,2,3 and 4:

* Participant involved in another interventional clinical study
* Person deprived of liberty by judicial order
* Person under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Exploring PGI2 pathway in skin microvascular reactivity | Day 1
  Comparison of skin perfusion measured with laser speckle contrast imaging (LSCI) on the calf, and expressed as arbitrary perfusion units, in response to local cathodal current application, between the three groups

SECONDARY OUTCOMES:
Involvement of COX-1 and 2 in cutaneous current-induced vasodilation | Day 1
  1. Comparison of skin perfusion measured with LSCI on the calf, in response to local current application, during local infusion of ketorolac (COX-1 blocker), and meloxicam (COX-2 blocker), using skin microdialysis, between the three groups.
Involvement of sensory nerves in cutaneous current-induced vasodilation | Day 1
  2. Comparison of skin perfusion measured with LSCI on the calf, in response to local current application, after local infusion of lidocaine, between the three groups.
IP receptor function | Day 1
  3. Comparison of skin perfusion measured with LSCI on the calf, in response to intradermal infusion of treprostinil using skin microdialysis, between the three groups.
Involvement of NO et EETs pathways in cutaneous current-induced vasodilation | Day 1
  4. Comparison of skin perfusion measured with LSCI on the calf, in response to local current application, during local infusion of NG-Monomethyl-L-arginine (L-NMMA) and fluconazole using skin microdialysis, between the three groups.
Expression of different components of PGI2 pathway in the skin : PTGS1/2 | Day 1
  5. Comparison of the expression of Prostaglandin-Endoperoxide Synthase (PTGS1/2 (COX1/2)), in the skin of the calf, between the three groups and a fourth group of foot skin biopsies from patients with diabetes, neuropathy and DFU undergoing lower-limb surgery.
Expression of different components of PGI2 pathway in the skin : PTGIS | Day 1
  5. Comparison of the expression of PTGIS (CYP8A1) in the skin of the calf, between the three groups and a fourth group of foot skin biopsies from patients with diabetes, neuropathy and DFU undergoing lower-limb surgery.
Expression of different components of PGI2 pathway in the skin : PTGIR | Day 1
  5. Comparison of the expression of PTGIR (IP-receptor) in the skin of the calf, between the three groups and a fourth group of foot skin biopsies from patients with diabetes, neuropathy and DFU undergoing lower-limb surgery.
Expression of different components of PGI2 pathway in the skin : TBXA2R | Day 1
  5. Comparison of the expression of TXA2R (TP-receptor) in the skin of the calf, between the three groups and a fourth group of foot skin biopsies from patients with diabetes, neuropathy and DFU undergoing lower-limb surgery.
role of PGI2 pathway on cell migration in vitro | Day 1
  6. Cell migration observed on wounded 3D skin equivalents made from cells collected from the three groups and from a fourth group of patients undergoing lower-limb surgery. Fibroblasts and kératinocytes migration on 3D reconstructed skin models.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes Centre d'investigation clinique, Grenoble, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data sending an e-mail to : jlcracowski@chu-grenoble.fr or mroustit@chu-grenoble.fr
Supporting Information: Study Protocol

REFERENCES:
- [Background] Knebel SM, Sprague RS, Stephenson AH. Prostacyclin receptor expression on platelets of humans with type 2 diabetes is inversely correlated with hemoglobin A1c levels. Prostaglandins Other Lipid Mediat. 2015 Jan-Mar;116-117:131-5. doi: 10.1016/j.prostaglandins.2014.12.002. Epub 2015 Jan 21. PMID 25617843
- [Background] Gohin S, Sigaudo-Roussel D, Conjard-Duplany A, Dubourg L, Saumet JL, Fromy B. What can current stimulation tell us about the vascular function of endogenous prostacyclin in healthy rat skin in vivo? J Invest Dermatol. 2011 Jan;131(1):237-44. doi: 10.1038/jid.2010.267. Epub 2010 Sep 9. PMID 20827283
- [Background] Gibbons CH, Freeman R, Veves A. Diabetic neuropathy: a cross-sectional study of the relationships among tests of neurophysiology. Diabetes Care. 2010 Dec;33(12):2629-34. doi: 10.2337/dc10-0763. Epub 2010 Aug 30. PMID 20805259
- [Background] Hellmann M, Roustit M, Gaillard-Bigot F, Cracowski JL. Cutaneous iontophoresis of treprostinil, a prostacyclin analog, increases microvascular blood flux in diabetic malleolus area. Eur J Pharmacol. 2015 Jul 5;758:123-8. doi: 10.1016/j.ejphar.2015.03.066. Epub 2015 Apr 3. PMID 25843412